CLINICAL TRIAL: NCT04845646
Title: Phase I Open Label, Drug-Drug Interaction, Study to Evaluate the Effect of Itraconazole and Phenytoin on the Pharmacokinetics of ASC41 in Healthy Volunteers and A Study to Evaluate the PK, Safety and Tolerability in Subjects With Non-alcoholic Fatty Liver Disease (NAFLD).
Brief Title: DDI Study of ASC41 in HV and the PK, Safety and Tolerability in Subjects With NAFLD.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gannex Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASC41-105
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy; NAFLD
Keywords: Healthy; NAFLD; DDI (Drug-Drug Interaction); Itraconazole; Phenytoin; THR beta agonist; ASC41
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Itraconazole; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ASC41 + Itraconazole group (Experimental): 1. ASC41 5 mg po, One 5 mg ASC41 tablet on day 1 and 11.
  2. Itraconazole oral capsule 200 mg po qd (2 capsules given 1x/day or 200 mg/day) on days 6-16.
  Interventions: Drug: ASC41; Drug: Itraconazole
- ASC41 + Phenytoin group (Experimental): 1. ASC41 5 mg po, One 5 mg ASC41 tablet on day 1 and 19.
  2. Phenytoin oral capsule 300 mg (100 mg 3 x/day) on days 6-19.
  Interventions: Drug: ASC41; Drug: Phenytoin
- ASC41 group (Experimental): (1) ASC41 5 mg po. One 5 mg ASC41 tablet on day 1.
  Interventions: Drug: ASC41

INTERVENTIONS:
Drug: ASC41 — 5mg/tablet
Drug: Itraconazole — 200mg/capsule
  Arms: ASC41 + Itraconazole group
Drug: Phenytoin — 300mg/capsule
  Arms: ASC41 + Phenytoin group

SUMMARY:
The primary objective of this study is to evaluate the effect of itraconazole, a strong inhibitor)of cytochrome P4503A , and phenytoin a strong inducer of cytochrome P450 3A, CYP3A4, CYP1A2 and CYP2C19 on the pharmacokinetics of ASC41, a THR beta agonist tables in healthy subjects. The PK, Safety and Tolerability of ASC 41 in Subjects with NAFLD will also be evaluated. Approximately 24 subjects including 16 healthy volunteers (HVs) and 8 subjects with NAFLD will be enrolled. This study consists of 3 cohorts.

DETAILED DESCRIPTION:
This multiarm study in HVs and subjects with NAFLD is designed to further characterize the PK, safety and tolerability of ASC41. Part I of the study will assess the effect of itraconazole and phenytoin on the single-dose PK of ASC41 in HVs. Part II of the study will evaluate the PK, safety and tolerability of a single dose of ASC41 in subjects with NAFLD. The pharmacokinetics of ASC41 and its metabolite ASC41-A will be assessed in both parts I and II. The secondary objective of the study is to characterize the safety and tolerability of oral ASC41 in subjects in the U.S. with NAFLD and in HVs. Approximately 24 male and female participants will be enrolled. This study consists of 3 cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Part I Healthy subjects between 18 to 55 years of age
* Part II

  1. Subjects with NAFLD
  2. Subjects between 18 to 65 years of age

Key Exclusion criteria:

* Part I

  1. A history of thyroid disease
  2. A history of, or current liver disease, or liver injuries
  3. Platelet count <150,000/mcL
  4. INR> 1.2
  5. History of, or current electrocardiogram (ECG) abnormalities, arrhythmias or heart valve diseases judged to be clinically significant by the investigator
* Part II

  1. A history of thyroid disease
  2. Current or history of cirrhosis or decompensated liver disease
  3. AST or ALT > 5X ULN
  4. DBIL > ULN
  5. Acute or chronic liver disease other than NAFLD
  6. A history of bariatric surgery
  7. HbA1c >9.5% at screening
  8. Testosterone or estrogen replacement therapy
  9. Inducers or inhibitors of CYP3A4, including herbal therapies such as St John's Wort (CYP3A4 Inducer)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
AUC of ASC41 | Up to 24 days
  Evaluate the Area under the plasma concentration versus time curve.
Cmax of ASC41 | Up to 24 days
  Evaluate the Peak Plasma Concentration.

SECONDARY OUTCOMES:
t1/2 of ASC41 | Up to 24 days
  Evaluate the Terminal-Phase Half-Life.
CL/F of ASC41 | Up to 24 days
  Evaluate the Apparent Systemic Clearance.
Vd/F of ASC41 | Up to 24 days
  Evaluate the Apparent Volume of Distribution.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 24 days
  Occurrence of Serious Adverse Event (SAE), Adverse Event (AE) resulting in treatment discontinuation and/or dose reductions, and AE of special interest, from baseline up to 24 days.

CONTACTS AND LOCATIONS:
Locations (1):
- ICON early Phase Services LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided